CLINICAL TRIAL: NCT03193684
Title: Effect of Empagliflozin on Hepatic Glucose Metabolism: Role of Autonomic Nervous System
Brief Title: Empagliflozin and Hepatic Glucose Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC20170214H; 2R01DK097554-06 (NIH)
Record Dates: First submitted 2017-06-17; First posted 2017-06-21 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hepatic Glucose Metabolism
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: subjects will receive in parallel a treatment with empagliflozin or placebo for 3 months hepatic glucose metabolism and norepinephrine turnover will be studied before and after treatment
Who Masked: Participant, Investigator
Masking Description: the study is placebo controlled double blinded. randomization will be made by pharmacist and the randomization code will be kept in the pharmacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Experimental): empagliflozin 25 mg per day
  Interventions: Drug: Empagliflozin 25 MG
- control (Placebo Comparator): matching placebo 1 pill per day
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Empagliflozin 25 MG — subjects will receive daily dose of 25mg of empagliflozin for 3 months
  Arms: Treatment
Drug: Control — Placebo
  Other Names: Placebo
  Arms: control

SUMMARY:
the aim of this study is to examine the role of autonomic nervous system in the increase in hepatic glucose production in response to glucosuria caused by inhibition of renal glucose uptake

DETAILED DESCRIPTION:
Purpose/Objectives: To investigate the effect of empagliflozin, an SGLT2 inhibitor on hepatic glucose production and the role of autonomic nervous system in mediating the increase in hepatic glucose production in response glucosuria Research Design/Plan: the role of autonomic nervous system in the increase in hepatic glucose production caused by empagliflozin will be examined with norepinephrine (NE) turnover in two protocols. The first protocol is cross sectional, in which 36 T2DM patients will receive hepatic glucose production (HGP) and NE turnover will be measured before and after empagliflozin or placebo administration. In protocol 2, diabetic and non-diabetic subjects will receive baseline HGP, NE turnover, hepatic glucose uptake (HGU) and liver fat measurement before at 2 days after the start and 12 weeks after empagliflozin or placebo treatment.

Methods: the following techniques will be employed (1) Measurement of hepatic glucose production with 3H-glucose infusion, with and without glucose clamp, (2) substrate oxidation with indirect calorimetry and plasma ketone/lactate/insulin/glucagon concentrations; (3) Measurement of HGU with Oral-IV double tracer infusion; (4) Measurement of whole body norepinephrine turnover with 3H-norepinephrine infusion; (5) Measurement of heart rate variability; (6) Measurement of liver fat content with 1H-MRS Clinical Relevance: The results of the present studies will help identify the mechanism responsible for the increase in HGP caused by empagliflozin and the increase in ketone production. The first action of the drug ameliorates its clinical efficacy while the second increases the risk of adverse events (ketoacidosis). Identifying the mechanisms underlying these actions will help developing therapeutic strategies which increase the drug clinical efficacy and mitigates its adverse events.

ELIGIBILITY:
Inclusion Criteria:

* eGFR>60 ml/min healthy volunteers type 2 diabetes patients who otherwise healthy

Exclusion Criteria:

* eGFR <60 T2DM patients on insulin, GLP-1 RA or SGLT2 treatment Major organ disease type 1 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abdul-Ghani, MD, PhD, Principal Investigator — Diabetes Division, UTHSCSA
Locations (1):
- Diabetes Division, UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 36 | 36
Completed | 36 | 35
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (2) | 46 (2) | 51 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 18 | 19 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Effect of Empagliflozin on Autonomic Nervous System
Description: autonomic activity will be measured with as NE turnover rate.
  Total-body NE turnover rate was measured with 3H-NE infusion. A prime (3.8 µCi)-continuous (0.38 µCi/min) infusion of 3H-NE was started and continued for 60 minutes. Arterialized blood samples were collected before the start and between the 40-60 minute time period after the start of 3H-NE infusion. Total body NE turnover rate was calculated as the 3H-NE infusion rate (dpm/min) divided by the steady state plasma 3H-NE specific activity (dpm/pg) after 30 minutes
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: ng/min
Arm/Group | Treatment | Control
Number analyzed (Participants) | 36 | 36
ng/min
  Baseline NE Turnover | 480 (42) | 621 (87)
  12 weeks NE Turnover | 355 (52) | 635 (99)

2. Secondary Outcome: Hepatic Glucose Production
Description: HGP will be measured with tracer dilution technique
Time Frame: Baseline and 12 weeks
Population: one patient in treatment arm did not complete the study due to Covid-19.
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Treatment | Control
Number analyzed (Participants) | 24 | 12
mg/kg/min
  Baseline | 2.57 (0.15) | 2.63 (0.16)
  Week 12 | 3.15 (0.21) | 2.50 (0.15)

3. Other Pre Specified Outcome: Absolute Percentage Change From Baseline to 12 Weeks in Hepatic Fat Content
Description: the effect of treatment on hepatic fat content will be measured with MRS.
Time Frame: Baseline and12 weeks
Population: Thirty individuals with T2D and 27 without were randomly assigned to receive in double-blind fashion empagliflozin or matching placebo (2:1 ratio) for 12 weeks.
Measure: Mean (Standard Error); unit: percentage of liver fat content
Arm/Group | Treatment | Control
Number analyzed (Participants) | 30 | 27
percentage of liver fat content | -2.39 (0.79) | 0.91 (0.64)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 2/36 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=36) | Control (N=36)
Vaginal yeast infection (Reproductive system and breast disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03193684/Prot_SAP_000.pdf